CLINICAL TRIAL: NCT06436001
Title: Comparing BlueDop Vascular Expert to Ankle-Brachial Index in the Identification of Peripheral Vascular Disease in All-comers and Diabetic Patients
Brief Title: Comparing BlueDop Vascular Expert to Ankle-Brachial Index in the Identification of Peripheral Vascular Disease
Status: Completed | Type: Observational
Sponsor: Dakota Vascular (Other)
Responsible Party: Sponsor
Other Study IDs: BlueDop_DakotaVascular study; CIRBI Link: CR00555039 (Other: Advarra IRB)
Record Dates: First submitted 2024-05-24; First posted 2024-05-30 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: Peripheral Arterial Disease; Diabetes Mellitus
Keywords: peripheral arterial disease; ankle brachial index; arterial duplex; Doppler waveform
MeSH Terms: conditions — Peripheral Arterial Disease; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- BlueDop Vascular Expert: BlueDop Vascular Expert assessment vs Full Leg Arterial Duplex
- Ankle Brachial Index: ABI assessment verses Full Leg Arterial Duplex

SUMMARY:
To compare the screening capabilities of the BlueDop Vascular Expert (BVE) and ankle brachial index (ABI) in peripheral arterial disease for all-comer patients and those with diagnosed diabetes mellitus.

DETAILED DESCRIPTION:
This retrospective and prospective single-center study to compare the accuracy and screening capabilities of BVE and ABI with that of conventional Full Leg Arterial Duplex (FLAD) was performed at a private clinic in Sioux Falls, South Dakota, USA, with data collected from March 2023 to March 2024. Currently, BVE carries the European CE Mark but does not yet have FDA approval for use in the United States. This study was undertaken with local IRB approval.

Patients 18 years or older who presented to the center were consented to have BVE, ABI, and FLAD performed. BVE examination of lower extremity arteries were performed following the instruction for use (IFU). All examinations were performed by the same two registered vascular technologists. FLAD ultrasound was carried out with waveform interpretation interpreted by an outside cardiothoracic surgeon who specializes in treatment of arterial disease to determine the presence or absence of disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years or older who presented to the center were consented to have BVE, ABI, and FLAD performed.

Exclusion Criteria:

* Patients were excluded who had incomplete or inadequate data, if they were known to be currently pregnant, or if they had contraindications to Doppler ultrasound.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This retrospective and prospective single-center study to compare the accuracy and screening capabilities of BVE and ABI with that of conventional Full Leg Arterial Duplex (FLAD) was performed at a private clinic in Sioux Falls, South Dakota, USA, with data collected from March 2023 to March 2024.
Sampling Method: Non-Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
Sensitivity | data collected from March 2023 to March 2024
  Comparing ABI and BVE findings to FLAD
Specificity | data collected from March 2023 to March 2024
  Comparing ABI and BVE findings to FLAD
Accuracy | data collected from March 2023 to March 2024
  Comparing ABI and BVE findings to FLAD
Cohen's Kappa coefficient | data collected from March 2023 to March 2024
  Comparing ABI and BVE findings to FLAD

CONTACTS AND LOCATIONS:
Locations (1):
- Dakota Vascular, Sioux Falls, South Dakota, United States